CLINICAL TRIAL: NCT07025018
Title: A Multicenter, Randomized Controlled Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of HMPL-306 in Patients With Gliomas Harboring IDH1 and/or IDH2 Mutations
Brief Title: Phase I Study of HMPL-306 for the Treatment of Gliomas With IDH1 and/or IDH2 Mutations
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025-306-00CH1
Record Dates: First submitted 2025-05-28; First posted 2025-06-17 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Gliomas Harboring IDH1 and/or IDH2 Mutations
Keywords: gliomas; randomized controlled; Multicenter; IDH1 mutations; IDH2 mutations; safety run-in; MRI/MRS examination; Phase I; clinical study; pharmacokinetics (PK); pharmacodynamics (PD); efficacy; HMPL-306; perioperative study
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety run-in (Experimental): This phase plans to enroll patients with gliomas of IDH1 and/or IDH2 mutations. The DLT will be evaluated during the first 28 days after the initial dosage.
  Interventions: Drug: HMPL-306
- Perioperative study phase (Experimental): This phase plans to enroll patients with gliomas of definitive or suspected IDH1 and/or IDH2 mutations, who are scheduled for surgery. Patients who meet the inclusion criteria will be randomized to groups A, B, or C, to receive or not receive HMPL-306 treatment before surgery.
  Interventions: Drug: HMPL-306

INTERVENTIONS:
Drug: HMPL-306 — IDH small molecule inhibitor

SUMMARY:
This study is a multicenter, randomized controlled Phase I clinical study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of HMPL-306 in patients with gliomas harboring IDH1 and/or IDH2 mutations

DETAILED DESCRIPTION:
HMPL-306 is a dual IDH1/2 inhibitor. This is a multicenter, randomized controlled phase I clinical study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of HMPL-306 in patients with gliomas harboring IDH1 and/or IDH2 mutations.

The study consists of 2 parts: Part 1 (safety lead-in phase) and Part 2 (perioperative phase). Part 1 will determine safety and DLT. Part 2 will administer the HMPL-306 or no treatment to mIDH-positive gliomas.

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed about the study and voluntarily sign the informed consent form (ICF).
2. Age ≥ 18 years.
3. Safety Lead-In Phase: Patients with gliomas of a documented IDH1 and/or IDH2 mutation. Perioperative Study Phase: Patients with gliomas of definitive or suspected IDH1 and/or IDH2 mutations scheduled for surgery.
4. All patients must have at least one measurable lesion.
5. Karnofsky Performance Status (KPS) score ≥ 80% .
6. In the investigator's judgment, a life expectancy of ≥ 12 weeks.
7. Sufficient bone marrow and organ function.

Exclusion Criteria:

1. Previous treatment with IDH inhibitors.
2. Unresolved toxicity from previous antitumor treatments not reverted to ≤ Grade 1 (except for alopecia, skin pigmentation changes, and ≤ Grade 2 peripheral neuropathy).
3. Patients assessed by researchers to have high-risk or unstable conditions.
4. Having other malignancies or a history of other malignancies within 5 years prior to screening.
5. History of clinically significant liver disease, including active infection with viral hepatitis, or other active hepatitis, alcoholic liver disease, cirrhosis, etc.
6. Patients with HIV infection.
7. Pregnancy (positive pregnancy test before dosing) or currently breastfeeding women.
8. Presence of diseases or conditions affecting drug absorption.
9. Any other conditions, in the investigator's judgment, unsuitable for the study drug, will result in exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with Dose Limiting Toxicities (DLTs) | Up to 28 days after first dose of study drug
  DLT is defined as an adverse event (AE) that meets protocol defined DLT criteria during cycle 1 and is at least possibly related to study drug.
RP2D | From first dose of study drug to the time of progressive disease, assessed up to 24 months on average
  Determine the Phase II recommended dose (RP2D) of HMPL-306 in patients with gliomas harboring IDH1 and/or IDH2 mutations based on a comprehensive assessment.

SECONDARY OUTCOMES:
Maximum serum drug concentration | PK/PD weeks at screening through safety follow-up, assessed up to 24 months on average
  Blood samples will be obtained from all patients for determination of the maximum serum concentration of HMPL-306.
Time to maximum concentration | PK/PD weeks at screening through safety follow-up, assessed up to 24 months on average
  Blood samples will be obtained from all patients for determination time to maximum concentration of HMPL-306.
Area under the concentration-time curve (AUC) | PK/PD weeks at screening through safety follow-up, assessed up to 24 months on average
  Blood samples will be obtained from all patients for determination of the AUC of HMPL-306
Concentration of 2-HG in brain tumor tissue | PK/PD weeks at screening through safety follow-up, assessed up to 24 months on average
  Brain tumor tissue will be obtained from suitable patients for determination concentration of 2-HG.

OTHER OUTCOMES:
Objective Response Rate (ORR) | From first dose of study drug to the time of progressive disease, assessed up to 24 months on average
  ORR is defined as the proportion of subjects with confirmed best overall tumor response of Complete Response (CR) or Partial Response (PR) or Minor Response (MR).
Duration of response (DoR) | From first dose of study drug to the time of disease relapse or death, whichever comes first, assessed up to 24 months on average
  DoR defined as the time from the date of the first CR or PR or MR to the first date of progressive disease (PD) or death from any cause.
Progression-free Survival (PFS) | From first dose of study drug to the time of progressive disease or death due to any causes, whichever comes first, assessed up to 24 months
  PFS is defined as time from first dose date of study drug to date of progression or date of death from any cause, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Wu, Principal Investigator — Huashan Hospital; Bo Zhang, Study Director — Hutchmed
Locations (1):
- Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No